CLINICAL TRIAL: NCT04535323
Title: A Phase I, Single Arm, Prospective Study to Evaluate the Treatment of Genitourinary Syndrome of Menopause With Platelet Rich Plasma (PRP) in Women With a History of Breast Cancer
Brief Title: Platelet Rich Plasma for the Treatment of Genitourinary Syndrome of Menopause in Patients With Stage 0-III Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-002712; NCI-2021-02777 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Breast Adenocarcinoma; Genitourinary Syndrome of Menopause; Prognostic Stage 0 Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Carcinoma In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment of GSM (platelet rich plasma) (Experimental): Patients receive platelet rich plasma via injection into the vaginal area.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Biological: Therapeutic Autologous Platelet-rich Plasma

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Biological: Therapeutic Autologous Platelet-rich Plasma — Given via injection
  Other Names: PRP; Therapeutic PRP

SUMMARY:
This phase I trial is to find out possible benefits and/or side effects of platelet rich plasma for the treatment of genitourinary syndrome of menopause in patients with stage 0-III breast cancer. Platelet rich plasma is produced by collecting approximately 60-90 ml (4-6 tablespoons) of blood from the vein in patients' arm. The blood is spun using a centrifuge that separates the plasma and red blood cells. This allows doctors to collect the platelet rich plasma that is then loaded into individual, sterile syringes for injection. Giving platelet rich plasma may help relief symptoms of genitourinary syndrome of menopause in patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and feasibility of use of platelet rich plasma (PRP) treatment in breast cancer survivors with genitourinary syndrome of menopause (GSM).

SECONDARY OBJECTIVE:

I. To determine the preliminary efficacy in treatment of vaginal atrophy, urinary symptoms, assessment of sexual function, quality of life symptoms, and patient global impression of improvement and tolerability.

OUTLINE:

Patients receive platelet rich plasma via injection into the vaginal area.

After completion of study treatment, patients are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent or have an appropriate representative available to do so
* Ability to complete questionnaires by themselves or with assistance
* Ability to comply with treatment plan and follow-up visits
* Female patients >= 18 years
* Histological confirmation of adenocarcinoma of the breast stage 0 - III with no evidence of recurrence. Additionally, patients with stage III require three or more years from initial diagnosis with no evidence of recurrence.
* Natural, surgical, or medically induced menopause
* Self-report of vaginal itching, irritation, burning, dryness, or dyspareunia
* Triple negative or HER2 positive breast cancer =< 3 years from initial diagnosis

Exclusion Criteria:

* Receiving any form of hormone replacement therapy, including topical estrogens, testosterone, and dehydroepiandrosterone (DHEA) or selective estrogen receptor modulator (SERM), including tamoxifen and ospemifene in the previous 3 months prior to enrollment
* Personal history of vulvovaginal conditions such as lichen sclerosis, lichen planus, vulvovaginal condyloma, vaginal intraepithelial neoplasia, vaginal carcinoma, history of cervical or other gynecologic cancer, radical pelvic surgery, acute or recurrent urinary tract infection, genital infection, history of vaginal or pelvic radiation
* Chronic pelvic pain, current pelvic tension myalgia/muscle hypertonicity
* Pelvic organ prolapse greater than stage II
* Pelvic surgery within 6 months
* Known allergy to lidocaine or prilocaine
* Known allergy to silicone
* Use of vaginal moisturizers, lubricants, or homeopathic preparations within 2 weeks of therapy
* Hemoglobin < 11.6 g/dL or > 15.5 g/dL. If the laboratory reports a single, non-clinically significant result for any of these studies and is the only excluding factor it may be repeated 1 week later if the patient wishes. Normalization of that laboratory study will then be considered non-exclusionary
* Hematocrit < 34.9% or > 44.9%. If the laboratory reports a single, non-clinically significant result for any of these studies and is the only excluding factor it may be repeated 1 week later if the patient wishes. Normalization of that laboratory study will then be considered non-exclusionary
* White blood cell count < 3.4 X 10^9/L or > 10.5 X 10^9/L. If the laboratory reports a single, non-clinically significant result for any of these studies and is the only excluding factor it may be repeated 1 week later if the patient wishes. Normalization of that laboratory study will then be considered non-exclusionary
* Platelet count < 150 X 10^ 9/L or > 450 X 10^9/L. If the laboratory reports a single, non-clinically significant result for any of these studies and is the only excluding factor it may be repeated 1 week later if the patient wishes. Normalization of that laboratory study will then be considered non-exclusionary
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of the treatment
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy. NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 2 weeks post-treatment
  Safety endpoint is defined as a lack of serious adverse events. National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) will be used to grade the severity of adverse events that occur in this study.
Tolerability of planned injection regimen with pain scores | Up to 6 months post-treatment
  Feasibility will be based on whether or not 16 or more patients (> 80%) tolerate the planned injection regimen with pain scores during the procedure less than or equal to 4.

SECONDARY OUTCOMES:
Change in vaginal symptoms | Baseline up to 6 months
  Assessed using the vaginal assessment scale. Will be summarized using descriptive statistics.
Change in vulvar symptoms | Baseline up to 6 months
  Assessed using the vulvar assessment scale. Will be summarized using descriptive statistics.
Change in Day-to-Day Impact of Vaginal Aging score | Baseline up to 6 months
  Will be summarized using descriptive statistics.
Change in sexual function | Baseline up to 6 months
  Will assess change in Female Sexual Function Index score. Will be summarized using descriptive statistics.
Change in urinary symptoms | Baseline up to 6 months
  Assessed with Urogenital Distress Index 6 score. Will be summarized using descriptive statistics.
Objective vaginal changes - vaginal maturation index | Baseline up to 6 months
  Assessed with vaginal maturation index
Objective vaginal changes - vaginal health index score | Baseline up to 6 months
  Assessed with vaginal health index score
Objective vaginal changes - vaginal caliber | Baseline up to 6 months
  Assessed with vaginal caliber

CONTACTS AND LOCATIONS:
Overall Officials: Anita H. Chen, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Chen AH, Trabuco EC, Chumsri S, Thielen JM, Cornella JL, Shapiro SA, Heckman MG, Dukes RE, Arthurs JR, Blumenfeld SG, Yi J. Platelet-Rich Plasma for Genitourinary Syndrome of Menopause in Breast Cancer Survivors. Obstet Gynecol. 2025 Nov 1;146(5):728-736. doi: 10.1097/AOG.0000000000006081. Epub 2025 Sep 19. PMID 40966714
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials